CLINICAL TRIAL: NCT05455203
Title: The Development of a Brief Parent-Child Substance Use Educational Intervention for Black Families
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: On hold until funding is secured.
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000032674; R24DA051946 (NIH)
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Black parents and youth between the ages of 11-17 years from (n=40) parent-child dyads will be recruited for this study. The study is a formative qualitative study design with the intention of using findings for the adaptation and evidence-based intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADAPT-ITT guided implementation and adaptation (Experimental): ADAPT-ITT is an implementation science framework that guides the adaptation of evidence-based interventions (EBI) for specific settings or populations. ADAPT-ITT will be used to adapt the target interventions in partnership with a Family and Community Advisory Board, consisting of parents, caregivers, and leaders of family-based organizations in New Jersey.
  Interventions: Behavioral: ADAPT-ITT

INTERVENTIONS:
Behavioral: ADAPT-ITT — ADAPT-ITT is an implementation framework that guides adaptation of evidence-based interventions (EBI) for specific settings/populations. It will be used to adapt target interventions with a Family and Community Advisory Board. It has 8 phases: (1) Assess the risk profile of Black families in Paterson and East Orange, (2) Adopt or adapt an EBI, (3) Administer novel methods with families and children to facilitate the adaptation process, (4) Plan on what aspects of the EBI need to be adapted/how best to evaluate the adapted EBI, (5) Identify additional experts to assist in the adaptation process, (6) Integrate material from experts to adapt the EBI, (7) Train staff to implement the adapted intervention, and (8) Test the adapted intervention. Given time and financial constraints, five phases will be completed at the end of the pilot study. Qualitative data collected from individual dyad interviews will be used to inform the data.

SUMMARY:
The purpose of this study is to adapt a racial-specific parent-child substance use education intervention for Black families in Paterson and East Orange, New Jersey which can promote family bonding, communication, and supervision, as well as acknowledging racial and ethnic specific norms, values, and pride. The adaptation of this intervention will be designed based on the needs of Black parents and their children and direct input from them as stakeholders.

DETAILED DESCRIPTION:
The study is a formative qualitative study design with the intention of using findings for the adaptation and evidence-based intervention.

Study Approach: Using the ADAPT-ITT approach, we seek to first consult with Black families and stakeholders in cities that include a large population of Black people in Paterson and East Orange, New Jersey such as to understand their unique challenges in discussing substance use with their children while also seeking their guidance on the development of a racial specific substance use parent-child intervention. The investigator will use a proactive rather than a reactive approach to recruit study participants. A proactive approach brings project staff into direct contact with potential participants. This typically involves face-to-face contact with community leaders and organizations, as well as recruitment presentations and meetings in the community.

Aim 1: Collect qualitative data from Black parents and youth between the ages of 10-17 years from (n=20) parent-child dyads on the challenges, barriers, and facilitators to communicating about substance use. Recruitment will take place with partnership of community-based organizations and supportive family programs. Semi-structured interviews will be conducted with adolescents and their parents to solicit their perspectives on identifiable strategies that have worked to discuss substance use within their family, barriers and facilitators to effective prevention programs, and specific community and cultural norms regarding youth substance use. Interviews will be conducted separately where youth will be included in one focus group and interview and parents will be in a separate focus group and interview. This is done to allow for youth and parents to feel comfortable in sharing challenges pertaining to substance use prevention education.

Aim 2: Adapt a family and community-based substance use prevention intervention for Black youth and families in Paterson and East Orange, NJ. Using the ADAPT-ITT implementation framework, Phase 1 and 2 which include a family and community advisory board (consisting of three parent-child dyads and 3 community leaders) will be developed to guide the adaptation of the intervention. The proposed adapted intervention will build upon evidence-based parent-adolescent interventions such as the Strong African American Families-Teen (SAAF-T) and The Family Check Up.

Aim 2a: Phase 3 of ADAPT-ITT includes theater testing involving the family and community advisory board which will be responsible in reviewing the adapted interventions and providing feedback.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a Black/African American
* Children aged between 11-17
* Assent to being a part of the study
* Live in Paterson, New Jersey at the time of the study or Live in East Orange, NJ
* English as their first language.

Exclusion Criteria:

* Do not identify as Black/African American
* Do not assent to being a part of the study
* Does not live in Paterson, New Jersey or East Orange at the time of the study
* Does not read, speak or write in English

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Improving drug use communication between Black parents and children | 3 months
  Assessed using parent-child drug use communication scales. (This is a formative study that seeks to inform the intervention and the measures are being developed concurrently.)
Improving drug use communication between Black parents and children | 3 months
  Assessed using child drug use knowledge scale. (This is a formative study that seeks to inform the intervention and the measures are being developed concurrently.)

CONTACTS AND LOCATIONS:
Overall Officials: Ijeoma Opara, PhD LMSW MPH, Principal Investigator — Yale University
Locations (1):
- Oasis, Paterson, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No